CLINICAL TRIAL: NCT03468205
Title: The Relating Experienced To Recalled Breathlessness Observational Study
Acronym: RETRO
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Ekström, Associate Professor, Skane University Hospital
Other Study IDs: RETRO
Record Dates: First submitted 2018-02-26; First posted 2018-03-16 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Breathlessness; Dyspnea
Keywords: breathlessness; dyspnea; measurement
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main Cohort: Main cohort of patients meeting all of the eligibility criteria enrolled through newspaper adds, flyers and via non personal recruitment.
- Subgroup: Smaller group of patients, meeting eligibility criteria for the main study, enrolled through clinical visits. These patients will be followed more closely and also be recorded in a logbook in order for later review. Some of the participants in this group will be interviewed in a semi-qualitative interview about their experiences of breathlessness.

SUMMARY:
Background: Breathlessness is common through a range of chronic and life limiting diseases, such as chronic pulmonary disease and congestive hearth failure. There is a lack of knowledge concerning the understanding of the experience of breathlessness such as the relation between predicted, experienced and recalled breathlessness.

Method: Questions on breathlessness intensity will be asked to participants with breathlessness several times daily through a mobile application installed on the users own cellphone. The mean experienced breathlessness will be related to the predicted and the recalled breathlessness as well as to background factors.

DETAILED DESCRIPTION:
Background

Breathlessness, the subjective sensation of breathing discomfort, is common and appears with varying severity in daily life of people across a number of diseases such as congestive heart failure, asthma and chronic obstructive pulmonary disease (COPD). Breathlessness affects nearly a quarter of people 60+ and about half of patients with serious illness.[1-3] Breathlessness gives rise to increased anxiety and depression, increased risk of hospitalization and earlier death.[4]

Clinical care relies on the patient's history based on his/her symptom recall. The recalled level of recent breathlessness is used by the health professional in order to decide on the need for further investigations and treatment. Studies have shown that the recalled intensity of breathlessness during laboratory-provoked symptoms is not the same as the actually experienced symptom in daily life.[5] Further, studies has shown lacking communication in regards to breathlessness between doctor and patients.[7] Knowledge on how recalled intensity of breathlessness differs to the actual experienced intensity during activities of daily life is limited.

Several factors may influence the recalled symptom intensity including the highest and the final experienced intensity.[8, 9] A high intensity of breathlessness at the moment of recall has been correlated with higher recalled intensity than actually experienced during the period.[10] Also, even a very small decline in cognitive status was shown to influence the differences between recalled and experienced symptoms.[10]

Aims The primary aim is to evaluate the relationship between experienced breathlessness and 1) recalled (remembered) breathlessness; and 2) predicted future breathlessness. Secondary aims are to identify factors that influence the difference between experienced and recalled or predicted breathlessness, estimate the influence of breathlessness on physical activity.

Research questions.

Three types of breathlessness measures evaluated: experienced (at a time point), recalled (remembered) and predicted (future) breathlessness. The main research questions are:

1. How is the recalled breathlessness intensity for a time period (T1) related to:

   1.1. Experienced breathlessness intensity during T1 measured as:
   * Mean experienced intensity?
   * Peak experienced intensity?
   * Most recent experienced intensity
   * Perceived self-efficacy related to the breathlessness
   * Personality trait of high symptom sensitivity at baseline
   * Experienced trajectory of breathlessness (including constant; variable; increasing; decreasing; quick change) 1.2. Predicted breathlessness intensity for a future time period (T2)
2. How is the predicted breathlessness intensity for a subsequent time period (T2) related to:

   2.1 Experienced breathlessness intensity during T1? 2.2 Recalled breathlessness intensity during T1? 2.3 Experienced breathlessness intensity during T2?
3. Which factors are associated with the difference score between:

   3.1 Experienced and recalled breathlessness intensity during T1? 3.2 Predicted and experienced breathlessness intensity during T2?
4. Which breathlessness measures are related to physical activity prospectively measured during a time period (T2): [Clinical sub study]

   * Experienced intensity before T2?
   * Recalled intensity before T2?
   * The participant's predicted intensity of breathlessness for T2?
5. How do people think when they recall breathlessness over a defined time period (such as 'now', 'last 24 hours' and 'the last week')? [Clinical sub study]

Study procedures

Recruitment Potential participants will be identified by clinical and research staff at the centers of the participating investigators including primary care and internal medicine/cardiology departments in Blekinge, Örebro, and Skane University Hospital (Lund/Malmö). Participants will also be recruited through advertisements in national and local newspapers and magazines including those of the Swedish Respiratory Society, the Swedish Heart-Lung Foundation and the Heart-Lung Association, and on web-portals/sites.

Eligibility and Consent

Eligibility according to the inclusion and exclusion criteria, consent and study data are self-entered by the participant using an application on smart phone/pad.

Patients at the study centers who give their informed written consent will also be included in a clinical sub study, where additional data will be obtained on cognitive status, physical activity (using an activity monitor worn for one week), and from medical records, interview and registry follow-up.

Application based data collection

Baseline data will be recorded when starting the application and daily start and stop times will be set. At regular intervals during each day, the application will que the participant, using sound and homepage notifications, to self-rate the intensity of breathlessness during the last 10-15 minutes. Each que can be ignored or filled in at a later time. Recall of breathlessness during the preceding night or day and additional measurements are rated in the application each morning and evening, as well as for the whole week at the end of each week in the study. The participant can quit the application at any time and will be asked to complete the cessation/exit assessments for the completed part of the week. All application data, linked to the participant-specific study-ID, is encrypted and transferred to a central database in real time via the internet connection. If no Internet connection is available at the time of transfer or if for some reason the data transfer is interrupted, the data will be stored locally on the device and the application will try to resend when the connection is re-established and stabilized. The data will also be kept on the device until the end of the study to safeguard and create a redundancy. The database is located physically at Blekinge Institute of Technology and is used for several other clinical studies including Swedish National Study of Aging and Care in accordance with all relevant protocols for data security and integrity.

Clinical sub study

A subset of participants at the study centres will be asked to participate in a clinical sub study. In addition to the information regarding the main application-based study these participants will receive specific information about the sub study on paper and be asked to give their written informed consent to participate. A log of the study ID, Swedish social security number (for sub study patients only) is kept at each participating centre. Data including demographics, diagnoses, measures of pulmonary and cardiac function, treatments, and hospitalizations will be obtained from medical records and national registries with up to five years follow-up of diagnoses and hospitalizations (Patient Registry), dispensed medications (Prescribed Drug Registry) and survival (Causes of Death Registry). Participants will be asked to fill in a daily diary of the main events causing breathlessness and its impact during the day. Participants will also be invited to take part in a semi-qualitative interview focusing on their experience of breathlessness and specifically how they cognitively recall breathlessness over different time periods such as 'now', 'last 24 hours' or 'last week' using the study questionnaires and semi-structured qualitative interviews. This group of participants will also be interviewed shortly about their experiences on using the mobile application.

Power and Sample Size

To obtain a power of 80% to detect a clinically and statistically significant difference of 1 point on a 0-10 NRS between the mean experienced and the recalled daily breathlessness score, assuming a pooled standard deviation (SD) of 1.81, a minimum of 30 participants need to be included. This is consistent with the sample size of Meek et al.[11] To account for loss of data and ensure adequate power, at least 45 participants with data on 2 days or more will be included.

Ethical considerations

Informed consent to participate will be obtained from all participants, including that participation is entirely voluntary and does not affect care or clinical contacts and that participation can be discontinued at the discretion of the participant, and that upon discontinuing, no further data will be collected.

In the application, data are de-identified using a study ID number. For patients who do not participate in the clinical sub study, the Swedish social security number is not recorded. For patients in the clinical sub study, clinical data will be cross-linked with data collected through the application using a key between the study ID (used in the application) and the participant's Swedish social security number stored securely at the clinical centre.

Data will be presented on the group level only so that individual participants cannot be identified. The findings will be published in national and international peer-reviewed scientific journals. The de-identified data will be posted in open access data repository in accordance with the requirements of the scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-reported overall breathlessness intensity ≥ 3 on a 0-10 numerical rating scale (NRS) during the prior 2 weeks, that was not entirely caused by an acute infection such as a cold or pneumonia
* Able to walk without personal aid (rollator allowed)
* Can use a device (smart phone/pad) with Internet access regularly
* Ability to read and complete data entry at baseline
* Clinical stability with no expected need for hospital admission within one week
* Have not participated before in the present study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified by clinical and research staff at the centers of the participating investigators (see Research Team below) including primary care and internal medicine/cardiology departments in Blekinge, Örebro, and Skane University Hospital (Lund/Malmö). Participants will also be recruited through advertisements in national and local newspapers and magazines including those of the Swedish Respiratory Society, the Swedish Heart-Lung Foundation and the Heart-Lung Association, and on web-portals/sites, discussion forums and blogs.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Actual breathlessness. | Up to one week. Starting from installation of application.
  Intensity of breathlessness on a 0-10 Numerical Rating scale. 0 being no breathlessness and 10 being the worst imaginable breathlessness.

SECONDARY OUTCOMES:
Recalled breathlessness | Up to one week. Starting from installation of application.
  Intensity of breathlessness on a 0-10 numerical scale self. 0 being no breathlessness and 10 being the worst imaginable breathlessness.
Multidimensional dyspnea profile (MDP) | Up to one week. Starting from installation of application.
  Recording all dimensions of breathlessness
Predicted intensity of breathlessness on a 0-10 numerical rating scale | Up to one week. Starting from installation of application.
  Predicting future symptom level. 0 being no breathlessness and 10 being the worst imaginable breathlessness.
Perceived self-efficacy regarding breathlessness | Up to one week. Starting from installation of application.
  Rating on a 0-10 numerical rating scale. 0 being complete control of symptoms and 10 being the no control of symptoms..

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sandberg, MD, Study Director — Blekinge County Council Hospital
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gronseth R, Vollmer WM, Hardie JA, Olafsdottir IS, Lamprecht B, Buist AS, Gnatiuc L, Gulsvik A, Johannessen A, Enright P. Predictors of dyspnoea prevalence: results from the BOLD study. Eur Respir J. 2014 Jun;43(6):1610-20. doi: 10.1183/09031936.00036813. Epub 2013 Oct 31. PMID 24176991
- [Background] Lopez Varela MV, Montes de Oca M, Halbert RJ, Muino A, Perez-Padilla R, Talamo C, Jardim JR, Valdivia G, Pertuze J, Moreno D, Menezes AM; PLATINO Team. Sex-related differences in COPD in five Latin American cities: the PLATINO study. Eur Respir J. 2010 Nov;36(5):1034-41. doi: 10.1183/09031936.00165409. Epub 2010 Apr 8. PMID 20378599
- [Background] Bowden JA, To TH, Abernethy AP, Currow DC. Predictors of chronic breathlessness: a large population study. BMC Public Health. 2011 Jan 12;11:33. doi: 10.1186/1471-2458-11-33. PMID 21226957
- [Background] Lansing RW, Gracely RH, Banzett RB. The multiple dimensions of dyspnea: review and hypotheses. Respir Physiol Neurobiol. 2009 May 30;167(1):53-60. doi: 10.1016/j.resp.2008.07.012. Epub 2008 Jul 25. PMID 18706531
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Laviolette L, Laveneziana P; ERS Research Seminar Faculty. Dyspnoea: a multidimensional and multidisciplinary approach. Eur Respir J. 2014 Jun;43(6):1750-62. doi: 10.1183/09031936.00092613. Epub 2014 Feb 13. PMID 24525437
- [Background] Mead J. Dysanapsis in normal lungs assessed by the relationship between maximal flow, static recoil, and vital capacity. Am Rev Respir Dis. 1980 Feb;121(2):339-42. doi: 10.1164/arrd.1980.121.2.339. PMID 7362140
- [Background] Williams M, Garrard A, Cafarella P, Petkov J, Frith P. Quality of recalled dyspnoea is different from exercise-induced dyspnoea: an experimental study. Aust J Physiother. 2009;55(3):177-83. doi: 10.1016/s0004-9514(09)70078-9. PMID 19681739
- [Background] Walentynowicz M, Bogaerts K, Van Diest I, Raes F, Van den Bergh O. Was it so bad? The role of retrospective memory in symptom reporting. Health Psychol. 2015 Dec;34(12):1166-74. doi: 10.1037/hea0000222. Epub 2015 May 25. PMID 26010720
- [Background] Miravitlles M, Ferrer J, Baro E, Lleonart M, Galera J. Differences between physician and patient in the perception of symptoms and their severity in COPD. Respir Med. 2013 Dec;107(12):1977-85. doi: 10.1016/j.rmed.2013.06.019. Epub 2013 Jul 24. PMID 23890959
- [Background] Meek PM, Lareau SC, Anderson D. Memory for symptoms in COPD patients: how accurate are their reports? Eur Respir J. 2001 Sep;18(3):474-81. doi: 10.1183/09031936.01.00083501. PMID 11589344
- [Derived] Elmberg V, Ekstrom M. Effect of the trajectory of exertional breathlessness on symptom recall and anticipation: A randomized controlled trial. PLoS One. 2020 Sep 11;15(9):e0238937. doi: 10.1371/journal.pone.0238937. eCollection 2020. PMID 32915891
- [Derived] Sandberg J, Lansing R, Anderberg P, Currow D, Sundh J, Ahmadi Z, Palmqvist S, Ekstrom M. Relating Experienced To Recalled breathlessness Observational (RETRO) study: a prospective study using a mobile phone application. BMJ Open Respir Res. 2019 Feb 12;6(1):e000370. doi: 10.1136/bmjresp-2018-000370. eCollection 2019. PMID 30956800